CLINICAL TRIAL: NCT01353820
Title: Proof of Concept -Effects of Lactobacillus Delbruckii Lactis DN111244 Fermented Milk Consumption on Plasma Lipids Levels in Hypercholesterolaemic Adults.
Brief Title: Effects of Lactobacillus Delbruckii Lactis DN111244 Fermented Milk Consumption on Plasma Lipids Levels in Hypercholesterolaemic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU280
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hypercholesterolemia
Keywords: Midly hypercholesterolemic subjects; Probiotic; Cholesterol lowering; Dairy
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Active Comparator)
  Interventions: Dietary Supplement: 1- Low fat drinkable fermented by Lactobacillus Delbruckii lactis (DN111244) - >10E8 <5.10E9 cfu/mL
- 2 = Control product (Sham Comparator)
  Interventions: Dietary Supplement: 2- Low fat drinkable fermented by S. thermophilus and L. bulgaricus

INTERVENTIONS:
Dietary Supplement: 1- Low fat drinkable fermented by Lactobacillus Delbruckii lactis (DN111244) - >10E8 <5.10E9 cfu/mL — 1- Intervention with test product ( >10E8 to <5.10E9 cfu/ml of L. delbruckii lactis )
  Arms: 1 = Tested product
Dietary Supplement: 2- Low fat drinkable fermented by S. thermophilus and L. bulgaricus — 2- Intervention with control product
  Arms: 2 = Control product

SUMMARY:
The objective of this study is to investigate the effect of Lactobacillus Delbruckii lactis (DN111244) fermented milk consumption on relative change of plasma LDL-cholesterol concentration in hypercholesterolaemic adults after 8 weeks of product consumption versus control product.

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 18-75 years;
* BMI between 19 and 30 kg/m2,
* LDL-cholesterol plasma level between 130 mg/dL to 190 mg/dL (bounds included) with or without statin monotherapy,
* stabilized hypercholesterolemia (since more than 3 months),
* accepting to follow the dietary recommendations advisable for hypercholesterolemic patient (NCEP-ATP III guidelines),
* used to consume dairy products,
* for female: effective contraceptive methods used,
* agreeing to a written informed consent

Exclusion Criteria:

* plasma triglycerides (TG) levels > 350 mg/dL (4 mmol//L),
* any cardiovascular event (infarction, angina, surgical or endocoronary intervention, stroke, peripheral arteriosclerosis, etc) in the last 6 months,
* known allergy or hypersensitivity to milk proteins,
* systemic treatment or topical treatment likely to interfere with evaluation of the study parameters,
* subject currently involved in a clinical trial or in an exclusion period following participation in another clinical tria,
* subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject,
* diabetic subjects (type I and type II),
* any kind of disease likely to interfere with the evaluation of efficiency or safety of the product,
* for female subject: pregnancy, breast feeding or intention to become pregnant during the study,
* for female subject: subject likely to change her contraceptive method during the study,
* active heavy cigarette smokers (reported more than 20 cigarettes / day),
* subjects who are actively participating in a weight loss program or have participated in a weight loss program in the three months prior to screening for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AMED s.r.o (Poliklinika Budějovická), Prague, Czechia